CLINICAL TRIAL: NCT04707833
Title: Protocol for the Collection of Clinical Samples for Evaluation and Implementation of Serological Techniques for Screening for COVID-19 Infection at the University Hospital of Rouen
Brief Title: Evaluation of Serological Techniques for Screening for COVID-19 Infection at the University Hospital of Rouen
Acronym: SeroCOV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020/0126/HP
Record Dates: First submitted 2020-12-29; First posted 2021-01-13 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Corona Virus Infection
MeSH Terms: conditions — Coronavirus Infections | interventions — COVID-19 Serological Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient infected or cured from covid19 (Experimental): * Patients with an acute SARS-CoV-2 infection confirmed by a positive RT-PCR, hospitalized in COVID units or in COVID resuscitations,
  * Nurses at the Rouen University Hospital infected with COVID 19, and cured,
  * Patients with a high suggestive clinic for COVID-19 infection but with negative COVID-19 RT-PCR
  Interventions: Diagnostic Test: Serological testing for COVID-19 infection

INTERVENTIONS:
Diagnostic Test: Serological testing for COVID-19 infection — The tests used will be the following:
  EUROIMMUN SARS-CoV-2(IgA) ELISA ELISA SARS-CoV-2 (IgG) EUROIMMUN WANTAI SARS-CoV-2 Ab ELISA WANTAI SARS-CoV-2 IgM ELISA Abbott Architect SARS-CoV-2 IgG Diasorin SARS LINK CoV-2 S1/S2 IgG Roche ECL anti-SARS-Cov-2 (combined IgG IgM IgA)

SUMMARY:
At present, the offer of tests for the serological diagnosis of CoVID-19 (detection of IgG, IgM or IgA antibodies against CoV-2 SARS) is plethoric and is based on the use of a very large number of rapid diagnostic unit tests, a few dedicated high throughput automated systems or reagents on existing open systems. The offer will continue to expand in the coming months.

In order to meet the objectives mentioned by the Prime Minister, and confirmed in the HAS report of April 16, 2020 and in the opinion n°6 of the COVID-19 scientific council concerning the potential use of these serological tests at the end of the COVID-19 epidemic, the Virology laboratory wishes to validate the sensitivity and specificity of the tests it intends to use.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria in the retrospective "Negative/Potentially Interfering" group are as follows :

* Adult patient sampled prior to the onset of the COVID-19 epidemic (before January 2020)
* Patient presenting a coronavirus infection other than SARS-CoV-2, or other respiratory viral infections (influenza, metapneumovirus)
* Patients for whom a serum is kept in the biocollection declared under the number AC-2014-2293 and kept in the Institute of Clinical Biology, University Hospital of Rouen.

The criteria for inclusion in the "acute point infection" group are as follows:

* Patients screened by a positive RT-PCR for an SARS-CoV-2 infection
* Patients aged ≥ 18 years old
* Patients taken in charge in the emergency room / in a unit / in COVID resuscitation at the Rouen University Hospital.
* Patients having read and understood the briefing note
* Non-opposition to participation in the study

The criteria for inclusion in the "Sequential acute infection" group are as follows:

* Patients with positive RT-PCR for CoV-2-SARS infection
* Patients aged ≥ 18 years old
* Taken care of in a COVID unit at the Rouen University Hospital
* Having read and understood the briefing note and signed the informed consent form

The criteria for inclusion in the "Convalescent" group are as follows:

* Caregivers working at the UH of Rouen
* Screened by positive RT-PCR for SARS-CoV-2 infection,
* Healed for at least one month at the time of inclusion
* Having read and understood the briefing note and signed the informed consent form

Exclusion Criteria:

* Minor person
* Known Pregnancy
* Person deprived of liberty by an administrative or judicial decision or person placed under judicial protection / subtutorship or guardianship
* Person not affiliated with social security
* Person who does not understand and speak French

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2020-11-26 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of immunological Abbott Architect SARS-CoV-2 IgG Assay | 24 months
  Measurement of antibodies against COVID-19 infection (Sensitivity and specificity )

SECONDARY OUTCOMES:
Evaluation of immunological of EUROIMMUN SARS-CoV-2(IgA) ELISA, EUROIMMUN SARS-CoV-2 (IgG) ELISA, WANTAI SARS-CoV-2 Ab ELISA, WANTAI SARS-CoV-2 IgM ELISA, Diasorin LIAISON SARS CoV-2 S1/S2 IgG, Roche ECL anti-SARS-Cov-2 (combined IgG IgA) | 24 months
  Measurement of antibodies against COVID-19 infection (Sensitivity and specificity )

CONTACTS AND LOCATIONS:
Locations (1):
- Rouen University Hospital, Rouen, France